CLINICAL TRIAL: NCT05707104
Title: Comparative Effects of Pilates and Plyometric Training on Physical Performance of Volleyball Players
Brief Title: Pilates and Plyometric Training on Physical Performance of Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/22/0430
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Volleyball Players
Keywords: Performance; Pilates; plyometric; volleyball; sprint
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises (Experimental): performing Pilates exercises three times per week for 6 weeks while maintaining their regular physical activity and nutritional plans.
  Interventions: Other: Pilates Exercises
- plyometric exercises (Experimental): performing plyometric exercises three times per week for 6 weeks while maintaining their regular physical activity and nutritional plans.
  Interventions: Other: plyometrics exercises

INTERVENTIONS:
Other: Pilates Exercises — NO. Exercises Targeted muscles Repetitions
  1. Pelvic curl Abdominals, Hamstrings & Quadriceps Femoris, Gluteus Maximums. 05
  2. Chest lift Rectus Abdominus, Internal & External Oblique Muscles 10
  3. Leg lift supine Quadriceps Femoris, Internal & External Oblique Muscles 10
  4. Leg lift side Quadriceps Femoris, Posterior Spinal Group, Internal & External Oblique Muscle 10
  5. Leg full side Adductor Longus Brevis, Magnus , gracilis, Pectineus, muscles 10
  6. Spine twist supine Abdominals,Quadriceps & Hamstring group of Muscles 10
  7. Chest lift with rotation Internal & External Oblique, Rectus & Transverses Abdominus Muscles 5 on each side
  8. Back extension BACK EXTENSION Abdominal group, Gluteus Maximus & Hamstrings Muscle 5 each side Rest between exercises 20 seconds Rest between set of exercises 45 to 60 seconds
  Arms: Pilates exercises
Other: plyometrics exercises — 1. SIDE TO SIDE ANKLE HOPS STANDING JUMP AND REACH FRONT CONE HOPS 2×15 2×15 5×6
  2. SIDE TO SIDE ANKLE HOPS STANDING JUMP LATERAL JUMP BARRIER 2×15 5×6 2×15
  3. DOUBLE LEG HOPS LATERAL CONE HOPS 5×8 2×12
  4. DIAGONAL CONE HOPS LATERAL SPRINT 4×8 4×8
  5. LATERAL CONE HOPS SINGLE LEG BOUNDING LATERAL JUMP SINGLE LEG 4×12 4×7 4×7
  6. DIAGONAL CONE HOPS HEXAGONAL DRILL CONE HOPS WITH CHANGE OF DIRECTION SPRINT DOUBLE LEG HOPS LATERAL JUMP SINGLE LEG 2×12 2×12 4×6 3×8 4×6
  Arms: plyometric exercises

SUMMARY:
Volleyball is one of the famous games which is used in order to enhance and increase physical and game oriented skills in athletes and players. The main goal of athletic training and sports participation is to enhance athletic performance. Different types of training regimes (Pilates and Plyometric) are used on athletes to increase their physical performance. As volleyball is the game of power agility as well as speed. Physical fitness is one of the important parameters of this game. So, Pilates training strengthens the deep core muscles and improves movement, efficiency and muscle control. And plyometric training is to increase the power of subsequent movements using both natural elastic components of muscle and tendon and the stretch reflex. The aim of this study is to compare the effects of Pilates and Plyometric, on physical performance of volleyball players.

DETAILED DESCRIPTION:
This will be a Randomized Clinical Trial that will be conducted at Pakistan Sports Board and Coaching Centre, Lahore. Participants of the study are 38 that will be randomly allocated into 2 groups. The group A will perform Pilates three times per week for 6 weeks and group B will follow Plyometric training three times per week for 6 weeks. Participants of both groups will follow their regular warm up regime and nutrition plans. All participants will undergo a pre and post treatment test via Functional movement's screen test (FMST), vertical-jump test (VJT), 30m sprint test, sit and reach test. The data will be analyzed via SPSS version 21.

Key Words: Performance; Pilates; plyometric; sprint; volleyballVolleyball is one of the famous games which is used in order to enhance and increase physical and game oriented skills in athletes and players. The main goal of athletic training and sports participation is to enhance athletic performance. Different types of training regimes (Pilates and Plyometric) are used on athletes to increase their physical performance. As volleyball is the game of power agility as well as speed. Physical fitness is one of the important parameters of this game. So, Pilates training strengthens the deep core muscles and improves movement, efficiency and muscle control. And plyometric training is to increase the power of subsequent movements using both natural elastic components of muscle and tendon and the stretch reflex. The aim of this study is to compare the effects of Pilates and Plyometric, on physical performance of volleyball players.

This will be a Randomized Clinical Trial that will be conducted at Pakistan Sports Board and Coaching Centre, Lahore. Participants of the study are 38 that will be randomly allocated into 2 groups. The group A will perform Pilates three times per week for 6 weeks and group B will follow Plyometric training three times per week for 6 weeks. Participants of both groups will follow their regular warm up regime and nutrition plans. All participants will undergo a pre and post treatment test via Functional movement's screen test (FMST), vertical-jump test (VJT), 30m sprint test, sit and reach test. The data will be analyzed via SPSS version 21.

Key Words: Performance; Pilates; plyometric; sprint; volleyball

ELIGIBILITY:
Inclusion Criteria:

* • Male and female volleyball players

  * Age group 18-30years.
  * Participants having an experience of at least 1 year.
  * Participants that are practicing for three or more times in a week

Exclusion Criteria:

* Athletes with any musculoskeletal injuries;

  * Athletes with any systemic illness;
  * Novice players
  * Any injury within one month
  * Players not willing to participate
  * Psychologically unstable
  * Elite/ International players.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Vertical jump test | 6 week
  The Vertical Jump test is designed to measure an applicant's lower body strength. The applicant then crouches and using the arms and legs jumps as high as possible extending the dominant arm. Upon reaching the top of the jump the applicant must tap the gauge "fins" to mark the jump height.
Sit and reach test | 6 weeks
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. It was initially described by Wells and Dillon in 1952 and is probably the mostly used flexibility test.
30m sprint test | 6 weeks
  The aim of this test is to determine acceleration and speed.The test involves running a single maximum sprint over 30 meters, with the time recorded.
ILLINOIS AGILITY TEST | 6 weeks
  The objective of this study is to monitor the athletes development in Agility. This test the subjects ability to turn in different directions and quickly change speeds. 37

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, phd, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No